CLINICAL TRIAL: NCT05731063
Title: Computer Guided Simultaneous Implant Placement With Tri-cortical Ridge Augmentation Using Chin Cortical Bone Struts in Anterior Atrophic Maxilla: A Case Series
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdrabelnaby Abdelrahman, Dentist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2722
Record Dates: First submitted 2022-11-14; First posted 2023-02-16 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Ridge Augmentation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ridge augmentation surgery (Other): Computer guided simultaneous implant placement with tri-cortical ridge augmentation using chin cortical bone struts in anterior atrophic maxilla
  Interventions: Procedure: Computer guided simultaneous implant placement with tri-cortical ridge augmentation using chin cortical bone struts

INTERVENTIONS:
Procedure: Computer guided simultaneous implant placement with tri-cortical ridge augmentation using chin cortical bone struts — fabrication of surgical guide to aid in chin bone harvesting and another guide to help for accurate placement and simultaneous placement in anterior maxillary defective area.

SUMMARY:
10 patients having deficient anterior maxilla will be recruited and a preoperative CBCT will be done to evaluate the vertical and horizontal dimensions of the intended alveolar ridge. pre-operative manufacturing of the digital surgical guides performed for Harvesting of the chin cortical bone struts from the symphysial area in the donor site and for Placement of the grafted cortical bone struts and the implant in the recipient site. Intra operatively the donor site (Chin) will be prepared to harvest autogenous bone from the chin aided by the patient's prefabricated bone harvesting guide. The recipient site (Maxillary anterior defect) will be prepared to receive the chin grafts. Grafts will be screwed in position and implants will be screwed in its preparation until it gains primary stability from basal bone, using the prefabricated bone fixation-implant placement guide. Any gaps will be filled with autogenous bone particulates from the chin. A healing tie base Abutment will be screwed into the implant through the third cortex.

Primary stability will be assessed using Osstell device. An immediate postoperative CBCT will be done and superimposed on the preoperative CBCT to measure accuracy of plan transfer to make sure the planning was followed accurately.

Follow up after 6 months and CBCT will be done for bone formation and density assessment and implant exposure for implant stability measurement-using osstell and removal Healing abutment and consecutive prosthetic loading.

ELIGIBILITY:
Inclusion Criteria:

* Patients with single or Multiple missing Maxillary Anterior Teeth with vertically and horizontally defective ridges having adequate soft tissue ample.
* Patients who gave their consent for this trial.
* Males and females will be included.

Exclusion Criteria:

* Patients on bisphosphonates or drugs altering bone metabolism, within 2 months before initiating the study.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Patients allergic to drugs used in the study.
* Patients having a history of a major medical condition (ASA 3,4)
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised patients.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Active infection or severe inflammation in the area intended for implant placement.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly followed.
* Referred only for implant placement or unable to attend a 5-year follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-27 (Actual); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Bone quality (change in bone density) | T0 before surgery, T1 immediately after surgery, T2 after 6 month
  Serial CBCT scans measuring change in bone density in grey value

SECONDARY OUTCOMES:
Bone quantity (bone formation "height and width") | T0 before surgery, T1 immediately after surgery, T2 after 6 month
  Serial CBCT scans (T0 before surgery, T1 immediately after surgery, T2 after 6 month) measuring bone quantity in mm
Implant stability | day of the surgery and at 6 month
  measure primary stability immediately after implant placement and in the second surgery using Osstell device (ISQ value of 1-100)
Accuracy of Plan Transfer | 1-3 days postoperatively
  Superimposition of preoperative digital plan and the immediate postoperative CBCT to assess the positional discrepancy of the graft between the digitally plan versus the actual postoperative position will be measured in millimeters three dimensionally (anteroposterior, vertical and lateral position).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt